CLINICAL TRIAL: NCT06456177
Title: Assessment of Nociception in Obstetric Patients During Epidural Analgesia
Brief Title: Nociception Monitoring During Epidural Analgesia
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Michael Grach, Director of outpatient pain medicine clinic, Carmel Medical Center
Other Study IDs: 0056-21-CMC
Record Dates: First submitted 2024-05-30; First posted 2024-06-13 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Pain Relief
Keywords: Epidural Analgesia; Visual Analogue Scale; Nociception Level Index

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Assessment of nociception in obstetric patients during epidural analgesia — Comparing nociception in obstetric patients during epidural analgesia, subjectively, by Visual analog scale and objectively by monitoring Nociception level Index

SUMMARY:
Introduction and aim: Nociception monitors have been used to assess pain management in anesthetized patients. The investigators set out to evaluate whether Nociception Level (NOL) monitor (PMD-200 monitor with NOL technology , (Medasense Biometrics Ltd. Ramat Gan, Israel) yields reliable readings during labor, and whether the derived NOL index will be associated with Visual analogue scale (VAS) subjective level of pain before and after the onset of epidural analgesia.

Methods:

Following approval by the intuitional review board No 0056-21-CMC, thirty parturients scheduled for epidural analgesia due to labor pains will be included in this prospective study, after informed consent for participation in the study will be obtained. NOL monitoring device will be connected to the subject finger. Epidural analgesia will be performed as per institutional standards. Data of VAS and NOL index will be collected once a minute. The association between VAS and NOL before and after the onset of adequate analgesia will be evaluated.

DETAILED DESCRIPTION:
Introduction:

Epidural analgesia is the most effective method of labor pain relief to this day. The lumbar epidural analgesia aims to induce a sensory block from T10 to L1, while at the same time facilitating the motor action of the lower limbs (L2-L5), thereby enabling the continued cooperation of the mother in the birth process.

Pain assessment is crucial for pain management and to date relies almost solely on subjective monitoring using self-assessment scales of the subject, which can be affected by personality, behavior, and psychological characteristics. Objective tools to measure pain have been developed. They rely on the changes in the balance between sympathetic and parasympathetic activity and include the heart rate variability, blood pressure, skin electrical conductivity and the vasomotor reflex and the electroencephalogram pupil. Nociception represents the integrated response to painful stimuli including the neural, hormonal and behavioral activity. Combination of multiple nociception-related parameters yielded stronger associations with the noxious stimuli compared with each parameter alone.

The PMD-200 monitor with NOL technology (Medasense Biometrics Ltd. Ramat Gan, Israel) is a novel, propriety, monitoring device based on a combination of nociception related physiological variables including heart rate, heart rate variability, photo-plethysmographic waveforms, skin conductance, and their time derivative. Based on a random forest model, the device generates the Nociception level (NOL) index, displayed as a scale from 0-100 with 0 representing no nociception and 100 representing extreme nociception. A NOL level of less than 25 arbitrary units is associated with adequate analgesia in patients under general anesthesia.

So far, the objective assessment of pain has been restricted mainly to patients who were under general anesthesia. Data in conscious patients is scant . The study design is to evaluate how nociception changes in the awake patients, and especially, how its changes following blockade of the painful stimuli. Study population parturients who will be scheduled to receive epidural analgesia for labor. This allow us to study the nociceptive level index during uterine contractions before and after the onset of epidural analgesia.

Methods:

Following approval by the intuitional review board No 0056-21-CMC, 30 parturients will be recruited and signed informed consent will be obtained.

Study protocol:

Visual analogue scale (VAS) will evaluated every 3-5 minutes and maximal NOL value within a 30 second interval will be recorded as the corresponding NOL value. Study duration will be up to 40 minutes following adequate pain relief. Total duration up to 60 minutes per parturient.

Epidural analgesia will be performed according to the protocol procedure in our institution (either sitting or lateral position with loss of resistance with either air or saline). Following insertion of an epidural catheter, a test dose of 40 mg of lidocaine will be injected to exclude spinal placement. 3 minutes later a bolus of 10 ml of 0.125% bupivacaine and 50 mcg fentanyl will be administered. VAS and NOL evaluation will proceed for up to 30 minutes after epidural analgesia commenced.

Definitions:

Baseline values (No pain relief values) are those collected before analgesia was achieved. Post epidural analgesia (Pain relief values) are those collected after the commencement of analgesia. That is after VAS dropped to 50% of highest baseline values Inadequate Epidural: Parturients who still had a VAS > 50% of BL VAS 20 minutes after epidural injection. They were treated conventionally to control pain either by additional injection of local anesthetic, a repeated epidural or other modes of pain relief. Once diagnosed as failed epidural further data was not collected.

Outcomes:

The effect of pain relief using neuroaxial epidural analgesia in awake patients with intermittent painful stimuli (uterine contractions) the association between VAS and NOL will be evaluated.

Data analysis The measurements will be divided according to the pain status: adequate pain relief and no pain relief. The NOL and VAS distribution while with and without pain relief will be presented with Box-plots and the mean, standard deviation, median, interquartile range (IQR) and range. For each woman, the difference between the mean VAS measured while having no pain relief and the mean VAS measured while having adequate pain relief will be calculated. The difference between the VAS score with and without pain relief was compared using Wilcoxon signed rank test. P<0.05 was considered statistically significant. The same analysis will be performed for NOL values (separately).

As each pain evaluation included both NOL and VAS values, a LOESS - Local Regression, which is a nonparametric technique that uses local weighted regression to fit a smooth curve through points in a scatter plot, will be performed. The LOESS purpose is to demonstrate the association between the VAS and the NOL.

In order to present the pain measurements along the time since the follow-up onset, a LOESS curves will be also performed. The statistical analysis and data management will be conducted using SAS 9.4 software (SAS Institute Inc., Cary, NC, USA.).

ELIGIBILITY:
Inclusion Criteria:

* Parturient
* Age between 20-45 years
* Present pregnancy istheir second
* Singleton births
* Under Epiduarl analgesia

Exclusion Criteria:

* Age younger than 20 years or older than 45 years
* First pregnancy
* Multiple birth

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women parturient , age between 20-45 years Present pregnancy is their second, Singleton births, third trimester of pregnancy, delivery conducted under Epiduarl analgesia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of pain relief using neuroaxial epidural analgesia in parturient by Visual Analog Scale (VAS) | 60 minutes
  The effect of pain relief using neuroaxial epidural analgesia in awake patients with intermittent painful stimuli (uterine contractions) by reporting the Visual Analog Scale (VAS) displayed as a scale from 1-10, with 0 representing no nociception and 10 representing extreme nociception, when higher scores mean a worse outcome
Evaluation of pain relief using neuroaxial epidural analgesia in parturient by Nociception Level (NOL) index | 60 minutes
  The effect of pain relief using neuroaxial epidural analgesia in awake patients with intermittent painful stimuli (uterine contractions) by monitoring the Nociception Level (NOL) index displayed as a scale from 0-100 with 0 representing no nociception and 100 representing extreme nociception, when higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Koos, Dr. MD, Study Chair — danako@clalit.org.il
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided